CLINICAL TRIAL: NCT05830188
Title: Feasibility, Acceptability, and Effectiveness of a Coping and Resilience Intervention in Adolescents in the Post-COVID-19 Era
Brief Title: A Coping and Resilience Intervention in Adolescents
Acronym: CERIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Okki Dhona Laksmita, Principal Investigator, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ceria2022
Record Dates: First submitted 2022-12-21; First posted 2023-04-26 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: COVID-19 Pandemic
Keywords: coping; COVID-19; health-related quality of life; PTSD symptoms; resilience; school-based intervention; social support
MeSH Terms: conditions — COVID-19 | interventions — Coping Skills

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CERIA (Experimental): Participants in the experimental group will receive six-weekly 45-60 minutes CERIA sessions in a classroom setting.
  Interventions: Behavioral: Coping and Resilience Intervention for Adolescents
- Control (Active Comparator): Printing materials for the CERIA sessions will be given to school counselors who provide school counseling programs in the control group. There will be no face-to-face meeting between the participants in the control group and the interventionist.
  Interventions: Other: Printing materials of Coping and Resilience Intervention for Adolescents

INTERVENTIONS:
Behavioral: Coping and Resilience Intervention for Adolescents — It is a school-based resilience enhancement program to help adolescents build skills of positive coping and social support to minimize negative coping and distress by sharing, identifying, and discussing their feelings, thoughts, and actions regarding problems and stressful events.
  Other Names: CERIA
  Arms: CERIA
Other: Printing materials of Coping and Resilience Intervention for Adolescents — Printing materials for the CERIA sessions will be given to school counselors who provide school counseling programs in the control group.
  Other Names: Printing materials of CERIA
  Arms: Control

SUMMARY:
The primary purpose of this study is to assess the feasibility and acceptability of a coping and resilience intervention for adolescents in school settings named CERIA, in the post-coronavirus disease 2019 or COVID-19 era. Whereas the secondary purpose of this study is to assess the effect of the intervention among adolescents on several outcomes, including posttraumatic stress disorder (PTSD) symptoms, defensive coping, courageous coping, social support, resilience, and health-related quality of life (HRQOL), in the post-COVID-19 era, at baseline or pre-test (one week before), right after/immediate effect or post-test (one week after), and one-month follow-up or short-term effect (one month after intervention).

The research questions in this study include the following:

* Is CERIA feasible for adolescents in the post-COVID-19 era?
* Is CERIA acceptable for adolescents in the post-COVID-19 era?
* What is the effect of CERIA on PTSD symptoms, defensive coping, courageous coping, social support, resilience, and HRQOL in adolescents in the experimental group compared to those in the control group in the post-COVID-19 era?
* Are there any differences in the mean scores of PTSD symptoms, defensive coping, courageous coping, social support, resilience, and HRQOL between the experimental and control groups at:
* one week before,
* one week after, and
* one month after CERIA?

Participants in the experimental group will be given six-weekly 45-60 minutes CERIA sessions, whereas participants in the control groups will be treated as active control. Researchers will compare the experimental and control groups to see the effect of the intervention (CERIA) to decrease the adolescents' PTSD symptoms and defensive coping and increase courageous coping, social support, resilience, and HRQOL at three different time points: one week before intervention, one week after intervention, and one month after the intervention.

DETAILED DESCRIPTION:
Content Validity for the Intervention (An Expert Panel)

The content validity for the CERIA is aimed to validate the appropriateness of CERIA by an expert panel. Panel members will be selected based on their educational expertise and experiences related to the study. The experts who will be invited to participate in the panel have to meet the following criteria: 1) have more than five years of clinical or research experience in psychoeducation, adolescents, and/or related field, 2) be willing to participate in the content validity study, and 3) be able to effectively communicate in either English or Indonesian language. Since this study will be conducted in the school setting, panel members can include university/ faculty members who have experience with the study topic, school counselors (teachers who are responsible for counseling programs in the school), assistant principal of student affairs (dean of students), and/or assistant principal of academic affairs and curriculum. School nurses will also be invited if any and if possible.

The sample size of a content validity study is related to a satisfactory content validation index (CVI) that is applied to assess the content validity of each item of the intervention protocol. In this study, the CVI will be adopted to identify the required sample size and level of consensus of the expert panel. As recommended, six experts are needed to reach a satisfactory CVI of 0.83 for each item on the content validity assessment form.

Content Validity Study Procedure

A formal invitation will be delivered via telephone or email to solicit eligible experts to participate in the study. Once the experts accept the invitation, a cover letter, and the content validity assessment form will be mailed to them. The cover letter consists of the purpose of the study, the selection criteria of the expert panel, detailed information on the assessment form (the CERIA intervention protocol), and instructions for rating each item. The assessment form includes several items associated with the CERIA intervention protocol, including the intervention content (rationale of the topic, intervention approach, therapeutic principle or components of the intervention activities per session), intervention design (duration of each session, number of intervention session in total, frequency of each session, length of intervention, setting, interventionist criteria, group participants), and components of the intervention manual (a guide book for educators and another guide book for participants). The rating of each item is based on a 4-point Likert scale (4= very appropriate, 3= appropriate, 2= inappropriate, and 1= very inappropriate). If the experts scored any of the items below a score of 3, they will be asked to provide comments or suggestions with relevant evidence and references to help the study further refine the intervention protocol.

Data Analysis for the Content Validity

The item-level CVI (I-CVI) and the scale-level (S-CVI) will be applied to evaluate the content validity of each of the items and the whole CERIA intervention protocol, respectively. The I-CVI will be calculated by counting the number of experts who rate the items as "appropriate" (a score of 3) or "very appropriate" (a score of 4) and dividing that number by the total number of experts. Whereas the S-CVI will be evaluated by calculating the average I-CVI across the items. A CVI of 0.80 or higher and 0.83 are considered satisfactory values for the S-CVI and I-CVI, respectively. Any item with a low CVI will be revised based on the experts' comments or suggestions until the CVI reaches the predefined satisfactory value.

School Sample and Recruitment

Investigators will use a CONSORT flow diagram to describe the phases of this study. A purposive sampling technique will be used in this study to specifically select two public junior high schools with more than 400 students each. Data regarding the number of students at each school will be updated (in the second semester of the new academic year 2022-2023). Briefing meetings will be used to inform principals of eligible schools about the study, prior to the issuing of invitations to participate. Following this, eligibility interviews with school principals will be used to ascertain the current strategies used to promote resilience within the schools. Investigators will send an invitation letter to the school principals along with the study's information and request written consent for school participation. In the event that a school does not respond to the invitation or declines to participate, the school recruitment process will be repeated, with the next identified eligible school invited to participate. The process will be continued until two schools have been recruited.

Random Allocation of Schools

The allocation of the schools to be either the intervention or control group will be conducted using simple randomization by one of our study team members. Schools, parents of students, and enrolled students will be blinded to study group allocation.

Student Recruitment

Parent-informed consent will be required for student participation. In order to optimize parental consent for child participation, investigators will share our study information with the school community through parents' or guardians' WhatsApp groups or other existing platforms. Distribution of parental consent will be conducted in selected classrooms in the schools. Every classroom in the schools has the same probability of being chosen. Using a random number function (in Microsoft Excel), investigators will select two classrooms from each grade level to distribute the parent-informed consent along and study information. Classrooms that have been selected should be agreed upon by the school principal and classroom teachers. Within the parent study statement, investigators will provide contact information so that they can reach out if they have any questions about the study.

On the first day of student recruitment, investigators will distribute the parental consent along with the PedsQLTM 4.0 Generic Core Scale parent proxy to the students in the selected classrooms in order to be signed by their parents or guardians at home. Parents or guardians who agree to participate in the study can sign the consent form and proceed to complete the PedsQLTM 4.0, Generic Core Scale parent proxy directly. Those who do not wish to participate may leave the parent proxy field blank. Whether they agree or disagree that their child should participate in the study, all of them must return the consent form and the PedsQLTM 4.0, Generic Core Scale parent proxy to the research team the following day. Parents or guardians who do not return the parental consent will be contacted through a phone call to provide verbal consent or non-consent for their child to participate. For those who provide verbal consent, replacement study information (with parental consent) will be provided by mail. Additionally, informed student consent for participation, or a student consent form, is required from each participant prior to the completion of student surveys at each point of data collection. Hence, for students whose parents or guardians have agreed and returned the parental consent form, investigators will request that they complete and return a signed consent form.

Sample Size

Investigators use the G*Power sample size calculator under an F test with an analysis of variance based on some criteria. First, an effect size of 0.3-0.4 (medium) is used. Second, investigators used a two-tailed hypothesis testing, with an α error probability of 0.05, and a power of 0.95. Third, the number of groups is 2 (intervention and control groups), and the number of measurements is 3 (pre-test, post-test, and follow-up). The sample size from the calculator yields 100 participants in total, plus a 10% attrition rate from the total participants. Hence, our study should include at least 110 participants that will be divided into intervention (n= 55) and control groups (n= 55).

Baseline Data Collection Procedure

On the same day of the student consent form distribution, students who agree to participate will be requested to complete a sociodemographic characteristic questionnaire and the six outcome measures. However, the completion of the six outcome measures will be conducted over a two-time period on the same day to avoid boredom among the participants. In the first period, a sociodemographic questionnaire, CRIES-13, MSPSS, CYRM-28, and PedsQLTM 4.0 Generic Core version will be completed. The JCS completion will be conducted later in the second period at a time agreed upon by the researcher and participants. For students who are unable to present during the data collection, an online version of the measures will be provided. All of the data will be collected by data collectors who are blinded to the group allocation.

Intervention Delivery

Students who agree to participate will be randomly grouped; one group consists of 5-10 students. Investigators will set a schedule for the intervention sessions for all of the groups. On the following week, when the first session of the intervention will begin, an interventionist will deliver the CERIA for 45-60 minutes in a classroom setting. The session will be assisted by two research assistants who are responsible for shifting the groups. Sessions 1-6 will be repeated using the same format. Intervention attendance lists for each session containing the names of participants will be provided. Adherence to the intervention session is defined as all participants following the protocol and receiving treatment as allocated. Each participant who is unable to attend one of the intervention sessions will be provided with an online version of the session material for the session they missed. The interventionist will ask them to read the material and practice the exercises at home so they can easily get into the next session.

Post-test and Follow-up Data Collection Procedure

In the last session of the intervention, investigators will conduct an additional 30-45 minutes for a focused-group discussion in order to collect the participants' views about CERIA. A questionnaire about the participants' perspectives will also be distributed. Data collection for the secondary outcomes one week after intervention and one month after intervention will be conducted using the same format as the baseline data collection.

Interventionist

Only health professionals with at least a baccalaureate nursing degree are qualified to conduct the intervention. Reading and understanding the intervention manual is required for those who intend to deliver the intervention. In this study, only one interventionist (the principal investigator) from the research team will deliver the intervention sessions.

Intervention Development

The foundations of the intervention development were based on the adolescent disaster survivor's resilience model. In the model, pathways to predict resilience were identified. First, PTSD symptoms and defensive coping as risk factors predicted resilience in a negative pathway directly and indirectly. Second, social support and courageous coping as protective factors predicted resilience in a positive pathway also directly and indirectly. And, third, there was an indirect effect of PTSD symptoms on resilience through defensive and courageous coping. Major impacts on resilience in the model had been demonstrated by the roles of coping variables where defensive and courageous coping acted as mediators and helped explain the indirect effects between PTSD symptoms and resilience. Defensive and courageous coping reflected cognitive appraisals used by individuals to evaluate stress. Defensive coping started out as a protective mechanism followed by social support, which caused defensive coping to transform into courageous coping. In this process, social support also performed a critical role to enhance resilience. Hence, the intervention component in this study will address the roles of risk (stress and negative coping) and protective (social support and positive coping) factors in the development of resilience and health-related quality of life related to the COVID-19 pandemic.

Plan for Data Management/ Analysis

The collected data will be analyzed using IBM SPSS for Windows version 26 and assumed a statistical significance level of p ≤ 0.05. Data consistency checks will be conducted to verify the reliability of the data collected. In case of missing data, several approaches will be used depending on which type of missing data is: missing completely at random, missing at random, or missing not at random. Investigators may employ complete case analysis to overcome the missing completely at random because this suggests investigators drop all cases if investigators have one or more values missing in any of the variables required for analysis. Multiple imputations can also be used; in each dataset, the missing values will be replaced by values that are randomly sampled from the predictive distribution of the observed data. This approach will provide valid results when the data are missing at random while avoiding the loss of power (sample size reduction). Alternatively, single imputation will be used by replacing a single value that best represents the mechanism of the missing value; this could be the mean of a normally distributed continuous variable, mode or median of a categorical variable, a predicted value of a regression equation, or the last/ best/ worst observation carried forward.

Data from the feasibility and acceptability (primary outcomes) will be analyzed quantitatively and qualitatively. Quantitative analysis which will be specified to descriptive statistics analysis will be applied for data regarding the time required to recruit target participants, participant recruitment, participant retention, participant attrition rates, participant compliance with the intervention, participant compliance and completeness of evaluation measures at pre-test, participant compliance and completeness of evaluation measures at post-test, and participant compliance and completeness of evaluation measures at follow-up.

Qualitative analysis will only be applied to primary outcomes data regarding the acceptability measure: participants' perspective on the intervention, an exit survey, and interventionist' perspective on the intervention). A focus group discussion (FGD) from a selected group of participants will be conducted and the FGD will be recorded using an encrypted digital audio recorder and will be transcribed verbatim. All data will be analyzed thematically using a Theoretical Framework Analysis (TFA) to guide the analysis. The TFA consists of seven component constructs: affective attitude, burden, perceived effectiveness, ethicality, intervention coherence, opportunity costs, and self-efficacy. Our research team will conduct the analysis with regular consensus meetings.

For the secondary outcomes, a generalized estimating equation framework will be used to analyze the matched cohort of students that participate in three-time point of assessments: pre-test, post-test, and follow-up surveys, and participants lost at follow-up, on baseline demographic characteristics (gender, ethnicity, and living arrangement) and the six outcomes (CRIES-13, JCS-defensive coping, JCS-courageous coping, MSPSS, CYRM-28, PedsQLTM 4.0 Generic Core version). Additionally, a linear mixed model with fixed- and random effects will be carried out for sensitivity analysis for all secondary outcomes using intention-to-treat principles, whereby multiple imputations were used to assess the sensitivity of the results to missing data under the missing at random (MAR) assumption for students that are lost to follow-up. The fixed effect will be applied to the treatment group (intervention vs. control) and prognostic variables (age, gender, ethnicity, and living arrangement). Whereas the random effect will be applied to schools to account for the clustering of responses within schools. This analysis is aimed to analyze data on the mean differences between all participants from experimental and control groups who completed the pre-test, post-test, and follow-up surveys for all secondary outcomes.

Interim Analysis and Stopping Guideline

During the study and subsequent follow-up data collection, investigators do not expect any issues that would be harmful to the participants. Investigators have no established termination criteria, and investigators do not plan to perform interim analyses before the follow-up data collection is completed.

ELIGIBILITY:
Inclusion Criteria:

* being aged 12-18 years old
* being enrolled in the participating public junior high schools in Yogyakarta
* voluntarily agreeing to participate by completing both the student-assent and parent-informed consent forms

Exclusion Criteria:

* individuals with mental retardation, psychosis, or any neurological disorders

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 110 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Feasibility Measure: Time required to recruit to target participants | From date of parent informed consent and student assent forms distribution until the date of consents qualification by the investigators, assessed up to 1 week.
  Assessment on the length of participants recruitment.
Feasibility Measure: Participant recruitment rate | From the date of the participant recruitment, assessed up to 1 week.
  Assessment on the process when potential participants are given information about the study to gauge their interest in and desire to participate as research subjects prior to being enrolled.
Feasibility Measure: Participant retention rate | From the date of the participant recruitment until the date of follow-up measurement, assessed up to 14 weeks.
  Assessment on the the method and techniques used to prevent participants in the study from withdrawing or dropping out.
Feasibility Measure: Participant attrition rate | From the date of the participant recruitment until the date of follow-up measurement, assessed up to 14 weeks.
  Assessment on the loss of study participants over time.
Feasibility Measure: Participant compliance with intervention | assessed up to 6 weeks
  Assessment on the participant compliance with CERIA sessions using an attendance list.
Feasibility Measure: Participant compliance and completeness of evaluation measures at pre-test | On the date of the pre-test, assessed up to 1 day.
  Assessment on the participant compliance and completeness of the evaluation measures (pre-test) using a checklist.
Feasibility Measure: Participant compliance and completeness of evaluation measures at post-test | On the date of the post-test, assessed up to 1 day.
  Assessment on the participant compliance and completeness of the evaluation measures (post-test) using a checklist.
Feasibility Measure: Participant compliance and completeness of evaluation measures at follow-up | On the date of the follow-up, assessed up to 1 day.
  Assessment on the participant compliance and completeness of the evaluation measures (follow-up) using a checklist.
Acceptability Measure: Participants' perspective on the intervention | On the date of the last session of CERIA, assessed up to 1 day.
  A 17-item questionnaire that measure participants' perspective on the intervention and a focused-group discussion (FGD) under the theoretical framework of acceptability (TFA) to assess prospective (i.e. experienced) and retrospective (i.e. experienced) acceptability from the participants. There will be 12 open-ended questions developed by researchers to guide the FGD. The FGD will only be conducted in one of the group of participants (10 students).
Acceptability Measure: An exit survey (participants' perspective on the intervention) | On the following day after the last session of CERIA, assessed up to 1 week.
  A 17-item questionnaire and the 12 open-ended questions about discontinuation of the study (only for students who discontinue to participate in the study, but at least attend 1 session of CERIA).
Acceptability Measure: Interventionist's perspective on the intervention | On the date of each sessions (session 1 to 6) of CERIA, assessed up to 6 weeks.
  An 8-item question that measures interventionist's perspective on the CERIA.
Acceptability Measure: Content validity for the intervention (an expert panel) | Assessed up to 8 weeks.
  An expert panel (6-8 experts) to evaluate the validity of the CERIA based on intervention appropriateness (intervention's content, design, components for each sessions, and evaluation). Each component has a four Likert-type option from 4= very appropriate, 3= appropriate, 2= inappropriate, and 1= very inappropriate. Experts who have any questions/comments/suggestions about CERIA can write them down on a rating form.

SECONDARY OUTCOMES:
Children's Revised Revised Impact of Event Scale (CRIES-13) | One week before intervention, one week after intervention, and one-month after intervention
  It is a child-friendly scale to measure PTSD reactions or symptoms that covers three sub-scales: intrusion (items 1, 4, 8, and 9), avoidance (items 2, 6, 7, and 10), and arousal (items 3, 5, 11, 12, and 13). All of the items are on a 4-point Likert type scale ranged from not at all = 0, rarely = 1, sometimes = 3, and often = 5. Higher scores indicate higher PTSD symptoms. If the sum of the scores on the intrusion and avoidance is 17 or more, then the probability of a child to have the PTSD symptoms is very high. CRIES-13 has satisfactory internal consistency reliability with Cronbach alpha coefficients are as follows: Intrusion = 0.70; Avoidance = 0.73; Arousal = 0.60; Total = 0.80. Examination of the scale in Indonesian adolescent population has been conducted in our pilot study with satisfactory results on its content validity index (item and scale levels), confirmatory factor analysis, and internal consistency reliability.
Jalowiec Coping Scale (JCS) | One week before intervention, one week after intervention, and one-month after intervention
  This coping scale has Part A (use) and Part B (effectiveness). Investigators will only use Part A. All of the answer options are rated on a Likert scale ranged from 0 to 3 to reflect the coping strategies that the individual frequently demonstrated; the degree of use of the coping strategy is rated as: 0= never used, 1= seldom used, 2= sometimes used, or 3= often used. It has eight sub-scales, consist of 10-item confrontive, 13-item evasive, 9-item optimistic, 4-item fatalistic, 5-item emotive, 7-item palliative, 5-item supportant, and 7-item self-reliant coping styles. Raw scores for each style are the sum of all items within a specific coping style; the mean scores derive from the summation of all items divided by the number of items within the specific coping style. Raw scores for overall items range from 0-180; the higher the scores indicates the higher use of the coping styles. The Indonesian version of the JCS has been validated in our previous studies.
Multidimensional Scale of Perceived Social Support (MSPSS) | One week before intervention, one week after intervention, and one-month after intervention
  It is a 12-item scale which measures three types of supports: family, friends, and significant others. Each of the support consists of four items which responded by 7 options from 1= very strongly disagree, 2= strongly disagree, 3= mildly disagree, 4= neutral, 5= mildly agree, 6= strongly agree, and 7= very strongly agree. The higher the scores, the higher the level of social support perceived. The scoring procedure is undertaken according to its sub-scales: family (items 3, 4, 8, and 11), friends (items 6, 7, 9, and 12), and significant others (items 1, 2, 5, and 10); sum across the items in each sub-scale and divide by 4. Or, it can be scored by the total scale; sum across the 12 items and divide by 12. The Indonesian version of the scale has performed good validity and reliability.
Child and Youth Resilience Measure 28 (CYRM-28) | One week before intervention, one week after intervention, and one-month after intervention
  It has three sub-scales: individual capacities/ resources (items 2, 8, 9, 11, 13, 14, 18, 21, and 23), relationships with primary caregivers (items 5, 6, 7, 12, 17, 24, and 26), and contextual factors that facilitate a sense of belonging (items 1, 3, 4, 10, 15, 16, 19, 20, 22, 25, 27, and 28). Certain questions in the survey provide insight into certain sub-scales. To score each sub-scale, simply sum responses to the relevant questions. Investigators had conducted a pilot study of the scale in 854 Indonesian adolescents during COVID-19 pandemic. Results showed that Cronbach's alpha coefficients for the total scale, individual capacities, relationships with primary caregiver, and contextual factors were 0.94, 0.83, 0.87, and 0.88, respectively.
Pediatric Quality of Life Inventory (PedsQLTM) 4.0 Generic Core youth version and parent proxy | One week before intervention, one week after intervention, and one-month after intervention
  It has two versions, youth self-report and parent proxy-report, each has 23 items divided into four domains: 8-item physical functioning, 5-item emotional functioning, 5-item social functioning, and 5-item school functioning. Each item is rated on a 5-Likert option: never = 0, almost never = 1, sometimes = 2, often = 3, and almost always = 4, with scoring interpretation should be converted to 0-100 indicating the higher score the higher HRQOL. An Indonesian version of the scale has been examined among children with cancer with satisfactory results. Our study also has done piloting the scale among 766 Indonesian adolescents during COVID-19 pandemic. The Cronbach's alpha and composite reliability coefficients for total scale and sub-scale in both versions were acceptable (>0.70). The ICC coefficients for total scale and each sub-scale between the self-report and proxy-report were adequate (>0.80).

CONTACTS AND LOCATIONS:
Overall Officials: Okki D Laksmita, MSc, Principal Investigator — School of Nursing, College of Nursing, Taipei Medical University
Locations (1):
- Okki Dhona Laksmita, Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Particular data will be shared: Individual participant data that underlie the results reported in this article, after identification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose. For example, for meta-analysis study.

REFERENCES:
- [Background] Allen, S. F., Pfefferbaum, B., Nitiéma, P., Pfefferbaum, R. L., Houston, J. B., McCarter, G. S., & Gray, S. R. (2016). Resilience and coping intervention with children and adolescents in at-risk neighborhoods. Journal of Loss and Trauma, 21(2), 85-98. doi:https://doi.org/10.1080/15325024.2015.1072014
- [Background] Beames JR, Li SH, Newby JM, Maston K, Christensen H, Werner-Seidler A. The upside: coping and psychological resilience in Australian adolescents during the COVID-19 pandemic. Child Adolesc Psychiatry Ment Health. 2021 Dec 18;15(1):77. doi: 10.1186/s13034-021-00432-z. PMID 34922575
- [Background] Bonardi O, Wang Y, Li K, Jiang X, Krishnan A, He C, Sun Y, Wu Y, Boruff JT, Markham S, Rice DB, Thombs-Vite I, Tasleem A, Santo TD, Yao A, Azar M, Agic B, Fahim C, Martin MS, Sockalingam S, Turecki G, Benedetti A, Thombs BD. Effects of COVID-19 Mental Health Interventions Among Children, Adolescents, and Adults Not Quarantined or Undergoing Treatment Due to COVID-19 Infection: A Systematic Review of Randomised Controlled Trials. Can J Psychiatry. 2022 May;67(5):336-350. doi: 10.1177/07067437211070648. Epub 2022 Mar 11. PMID 35275494
- [Background] Bridgland VME, Moeck EK, Green DM, Swain TL, Nayda DM, Matson LA, Hutchison NP, Takarangi MKT. Why the COVID-19 pandemic is a traumatic stressor. PLoS One. 2021 Jan 11;16(1):e0240146. doi: 10.1371/journal.pone.0240146. eCollection 2021. PMID 33428630
- [Background] Eldridge SM, Lancaster GA, Campbell MJ, Thabane L, Hopewell S, Coleman CL, Bond CM. Defining Feasibility and Pilot Studies in Preparation for Randomised Controlled Trials: Development of a Conceptual Framework. PLoS One. 2016 Mar 15;11(3):e0150205. doi: 10.1371/journal.pone.0150205. eCollection 2016. PMID 26978655
- [Background] Esserman D, Allore HG, Travison TG. The Method of Randomization for Cluster-Randomized Trials: Challenges of Including Patients with Multiple Chronic Conditions. Int J Stat Med Res. 2016 Jan 8;5(1):2-7. doi: 10.6000/1929-6029.2016.05.01.1. PMID 27478520
- [Background] Fenwick-Smith A, Dahlberg EE, Thompson SC. Systematic review of resilience-enhancing, universal, primary school-based mental health promotion programs. BMC Psychol. 2018 Jul 5;6(1):30. doi: 10.1186/s40359-018-0242-3. PMID 29976252
- [Background] Fox-Wasylyshyn SM, El-Masri MM. Handling missing data in self-report measures. Res Nurs Health. 2005 Dec;28(6):488-95. doi: 10.1002/nur.20100. PMID 16287052
- [Background] Giannopoulou I, Galinaki S, Kollintza E, Adamaki M, Kympouropoulos S, Alevyzakis E, Tsamakis K, Tsangaris I, Spandidos DA, Siafakas N, Zoumpourlis V, Rizos E. COVID-19 and post-traumatic stress disorder: The perfect 'storm' for mental health (Review). Exp Ther Med. 2021 Oct;22(4):1162. doi: 10.3892/etm.2021.10596. Epub 2021 Aug 11. PMID 34504607
- [Background] Haase JE. The adolescent resilience model as a guide to interventions. J Pediatr Oncol Nurs. 2004 Sep-Oct;21(5):289-99; discussion 300-4. doi: 10.1177/1043454204267922. PMID 15381798
- [Background] Haase, J. E. (2004b). Resilience. In S. J. P. T. S. Bredow (Ed.), Middle Range Theories: Application to Nursing Research (pp. 341-367). Philadelphia, USA: Lippincott Williams & Wilkins.
- [Background] Haase JE, Heiney SP, Ruccione KS, Stutzer C. Research triangulation to derive meaning-based quality-of-life theory: adolescent resilience model and instrument development. Int J Cancer Suppl. 1999;12:125-31. doi: 10.1002/(sici)1097-0215(1999)83:12+3.0.co;2-7. PMID 10679883
- [Background] Haase JE, Kintner EK, Monahan PO, Robb SL. The resilience in illness model, part 1: exploratory evaluation in adolescents and young adults with cancer. Cancer Nurs. 2014 May-Jun;37(3):E1-12. doi: 10.1097/NCC.0b013e31828941bb. PMID 23519038
- [Background] Haase JE, Kintner EK, Robb SL, Stump TE, Monahan PO, Phillips C, Stegenga KA, Burns DS. The Resilience in Illness Model Part 2: Confirmatory Evaluation in Adolescents and Young Adults With Cancer. Cancer Nurs. 2017 Nov/Dec;40(6):454-463. doi: 10.1097/NCC.0000000000000450. PMID 27984241
- [Background] Jalowiec, A. (2003). The Jalowiec Coping Scale. In O. L. S. C. Dilorio (Ed.), Measurement of nursing outcomes (2 ed., Vol. Self care and coping, pp. 71-87). New York: Springer.
- [Background] Jaycox LH, Langley AK, Stein BD, Wong M, Sharma P, Scott M, Schonlau M. Support for Students Exposed to Trauma: A Pilot Study. School Ment Health. 2009 Jun 1;1(2):49-60. doi: 10.1007/s12310-009-9007-8. PMID 20811511
- [Background] Karbasi, Z., & Eslami, P. (2022). Prevalence of post-traumatic stress disorder during the COVID-19 pandemic in children: a review and suggested solutions. Middle East Current Psychiatry, 29(1), 74. doi:https://doi.org/10.1186/s43045-022-00240-x
- [Background] Laksmita OD, Chung MH, Liao YM, Haase JE, Chang PC. Predictors of resilience among adolescent disaster survivors: A path analysis. J Adv Nurs. 2020 Aug;76(8):2060-2071. doi: 10.1111/jan.14396. Epub 2020 May 19. PMID 32301129
- [Background] Lazarus, R., & Folkman, S. (1984). Stress, appraisal, and coping. New York, NY: Springer.
- [Background] Lee, J. H., Nam, S. K., Kim, A.-R., Kim, B., Lee, M. Y., & Lee, S. M. (2013). Resilience: A meta-analytic approach. Journal of Counseling & Development, 91(3), 269-279. doi:https://doi.org/10.1002/j.1556-6676.2013.00095.x
- [Background] Luthar SS, Cicchetti D, Becker B. The construct of resilience: a critical evaluation and guidelines for future work. Child Dev. 2000 May-Jun;71(3):543-62. doi: 10.1111/1467-8624.00164. PMID 10953923
- [Background] Masten AS. Ordinary magic. Resilience processes in development. Am Psychol. 2001 Mar;56(3):227-38. doi: 10.1037//0003-066x.56.3.227. PMID 11315249
- [Background] Masten AS, Lucke CM, Nelson KM, Stallworthy IC. Resilience in Development and Psychopathology: Multisystem Perspectives. Annu Rev Clin Psychol. 2021 May 7;17:521-549. doi: 10.1146/annurev-clinpsy-081219-120307. Epub 2021 Feb 3. PMID 33534615
- [Background] Masten AS, Motti-Stefanidi F. Multisystem Resilience for Children and Youth in Disaster: Reflections in the Context of COVID-19. Advers Resil Sci. 2020;1(2):95-106. doi: 10.1007/s42844-020-00010-w. Epub 2020 Jun 25. PMID 32838305
- [Background] Mesman E, Vreeker A, Hillegers M. Resilience and mental health in children and adolescents: an update of the recent literature and future directions. Curr Opin Psychiatry. 2021 Nov 1;34(6):586-592. doi: 10.1097/YCO.0000000000000741. PMID 34433193
- [Background] Moher D, Schulz KF, Altman DG. The CONSORT statement: revised recommendations for improving the quality of reports of parallel-group randomised trials. Lancet. 2001 Apr 14;357(9263):1191-4. PMID 11323066
- [Background] O'Shea ER, Phillips KE, O'Shea KN, Roney LN. Preparing for the Impact of COVID-19 on the Mental Health of Youth. NASN Sch Nurse. 2022 Mar;37(2):64-69. doi: 10.1177/1942602X211052626. Epub 2021 Dec 10. PMID 34889126
- [Background] Pinto TM, Laurence PG, Macedo CR, Macedo EC. Resilience Programs for Children and Adolescents: A Systematic Review and Meta-Analysis. Front Psychol. 2021 Nov 22;12:754115. doi: 10.3389/fpsyg.2021.754115. eCollection 2021. PMID 34880812
- [Background] Ravens-Sieberer U, Kaman A, Erhart M, Devine J, Schlack R, Otto C. Impact of the COVID-19 pandemic on quality of life and mental health in children and adolescents in Germany. Eur Child Adolesc Psychiatry. 2022 Jun;31(6):879-889. doi: 10.1007/s00787-021-01726-5. Epub 2021 Jan 25. PMID 33492480
- [Background] Ronen, T. (2021). The Role of Coping Skills for Developing Resilience Among Children and Adolescents. In M. L. Kern & M. L. Wehmeyer (Eds.), The Palgrave Handbook of Positive Education (pp. 345-368). Cham: Springer International Publishing.
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 Statement: updated guidelines for reporting parallel group randomised trials. BMC Med. 2010 Mar 24;8:18. doi: 10.1186/1741-7015-8-18. PMID 20334633
- [Background] Sekhon M, Cartwright M, Francis JJ. Acceptability of healthcare interventions: an overview of reviews and development of a theoretical framework. BMC Health Serv Res. 2017 Jan 26;17(1):88. doi: 10.1186/s12913-017-2031-8. PMID 28126032
- [Background] Shanahan L, Steinhoff A, Bechtiger L, Murray AL, Nivette A, Hepp U, Ribeaud D, Eisner M. Emotional distress in young adults during the COVID-19 pandemic: evidence of risk and resilience from a longitudinal cohort study. Psychol Med. 2022 Apr;52(5):824-833. doi: 10.1017/S003329172000241X. Epub 2020 Jun 23. PMID 32571438
- [Background] Smith, P., Perrin, S., Dyregrov, A., & Yule, W. (2003). Principal components analysis of the impact of event scale with children in war. Personality and Individual Differences, 34(2), 315-322. doi:https://doi.org/10.1016/S0191-8869(02)00047-8
- [Background] Steinhardt M, Dolbier C. Evaluation of a resilience intervention to enhance coping strategies and protective factors and decrease symptomatology. J Am Coll Health. 2008 Jan-Feb;56(4):445-53. doi: 10.3200/JACH.56.44.445-454. PMID 18316290
- [Background] Tal-Saban M, Zaguri-Vittenberg S. Adolescents and Resilience: Factors Contributing to Health-Related Quality of Life during the COVID-19 Pandemic. Int J Environ Res Public Health. 2022 Mar 8;19(6):3157. doi: 10.3390/ijerph19063157. PMID 35328845
- [Background] Tasijawa, F. A., & Siagian, I. (2022). School-based interventions to improve adolescent resilience: A scoping review. Open Access Macedonian Journal of Medical Sciences, 10(F), 33-40. doi:https://doi.org/10.3889/oamjms.2022.8063
- [Background] Theberath M, Bauer D, Chen W, Salinas M, Mohabbat AB, Yang J, Chon TY, Bauer BA, Wahner-Roedler DL. Effects of COVID-19 pandemic on mental health of children and adolescents: A systematic review of survey studies. SAGE Open Med. 2022 Mar 30;10:20503121221086712. doi: 10.1177/20503121221086712. eCollection 2022. PMID 35371484
- [Background] Ungar, M., & Liebenberg, L. (2011). Assessing resilience across cultures using mixed methods: Construction of the Child and Youth Resilience Measure. Journal of Mixed Methods Research, 5(2), 126-149. doi:https://doi.org/10.1177/1558689811400607
- [Background] Varni JW, Seid M, Kurtin PS. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. Med Care. 2001 Aug;39(8):800-12. doi: 10.1097/00005650-200108000-00006. PMID 11468499
- [Background] VicHealth. (2015). Interventions to build resilience among young people: a literature review. Retrieved from https://www.vichealth.vic.gov.au/-/media/ResourceCentre/PublicationsandResources/Mental-health/Interventions-to-build-resilience-among-young-people.pdf?la=en&hash=52060B1A4407D7FDCB24945F32DF675B012385A4
- [Background] Waselewski EA, Waselewski ME, Chang T. Needs and Coping Behaviors of Youth in the U.S. During COVID-19. J Adolesc Health. 2020 Nov;67(5):649-652. doi: 10.1016/j.jadohealth.2020.07.043. Epub 2020 Sep 12. PMID 32933836
- [Background] Zhang C, Ye M, Fu Y, Yang M, Luo F, Yuan J, Tao Q. The Psychological Impact of the COVID-19 Pandemic on Teenagers in China. J Adolesc Health. 2020 Dec;67(6):747-755. doi: 10.1016/j.jadohealth.2020.08.026. Epub 2020 Oct 8. PMID 33041204
- [Background] Zimet, G. D., Dahlem, N. W., Zimet, S. G., & Farley, G. K. (1988). The Multidimensional Scale of Perceived Social Support. Journal of Personality Assessment, 52, 30-41. doi:https://doi.org/10.1207/s15327752jpa5201_2
- [Background] Laksmita OD, Chung MH, Shieh YY, Chang PC. Psychometric Validation of the Indonesian Version of Children's Revised Impact of Event Scale 13. Int J Environ Res Public Health. 2022 Dec 19;19(24):17069. doi: 10.3390/ijerph192417069. PMID 36554952
- [Background] Laksmita OD, Chung MH, Liao YM, Chang PC. Multidimensional Scale of Perceived Social Support in Indonesian adolescent disaster survivors: A psychometric evaluation. PLoS One. 2020 Mar 13;15(3):e0229958. doi: 10.1371/journal.pone.0229958. eCollection 2020. PMID 32168332
- [Background] Sitaresmi MN, Mostert S, Gundy CM, Sutaryo, Veerman AJ. Health-related quality of life assessment in Indonesian childhood acute lymphoblastic leukemia. Health Qual Life Outcomes. 2008 Nov 9;6:96. doi: 10.1186/1477-7525-6-96. PMID 18992169
- [Background] Polit DF, Beck CT, Owen SV. Is the CVI an acceptable indicator of content validity? Appraisal and recommendations. Res Nurs Health. 2007 Aug;30(4):459-67. doi: 10.1002/nur.20199. PMID 17654487
- [Background] Davis RS, Meiser-Stedman R, Afzal N, Devaney J, Halligan SL, Lofthouse K, Smith P, Stallard P, Ye S, Hiller RM. Systematic Review and Meta-analysis: Group-Based Interventions for Treating Posttraumatic Stress Symptoms in Children and Adolescents. J Am Acad Child Adolesc Psychiatry. 2023 Nov;62(11):1217-1232. doi: 10.1016/j.jaac.2023.02.013. Epub 2023 Mar 20. PMID 36948393